CLINICAL TRIAL: NCT05356585
Title: Circulating Tumor DNA to Monitor the Efficacy of Total Neoadjuvant Therapy for Rectal Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor already published research that was to be obtained from this study.
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: CASE9221
Record Dates: First submitted 2022-04-27; First posted 2022-05-02 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer; Rectal Cancer
Keywords: total neoadjuvant treatment; tumor-specific assay; Circulating Tumor DNA; ctDNA
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Formalin-fixed, paraffin embedded tissue from the patient's colonoscopy or flexible sigmoidoscopy in surgeon's office will be sent to Natera for Signatera assay creation after enrollment onto the study
  Blood will be collected in Ethylenediamine tetraacetic acid (EDTA) tubes and sent to Natera via shipping materials provided by Natera.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: SignateraTM assay — A customized tumor-informed ctDNA test that, after receiving the tumor tissue, examines whole exome sequencing of a biopsied tumor to find the somatic tumor-derived mutations. From those mutations, the 16 most clonal mutations are used to create a personal assay

SUMMARY:
The purpose of this study is to use the SignateraTm assay created from rectal tumor biopsies to monitor participants' blood for fragments of DNA shed by tumor cells. The tumor DNA fragments are referred to as circulating tumor DNA, or ctDNA for short.

DETAILED DESCRIPTION:
Rectal cancer tissue samples that were collected from participants' previous biopsies will be sent to Natera for Signatera assay creation after enrollment onto the study.

One 6 mL tube of blood will be obtained at baseline prior to initiation of treatment. Blood will also be obtained in two 6 tubes at the following points: 3-4 weeks into chemoradiation therapy (CRT), after CRT, after chemotherapy, after surgery for those who undergo resection, and during surveillance 3 months after surgery or at the end of treatment for one year after completion of TNT (total neoadjuvant therapy).

The primary objective of the study is to estimate the percentage of patients with positive ctDNA at the end of TNT .

The secondary objectives of the study include:

1. Estimating the change in ctDNA after chemoradiation and chemotherapy
2. Characterize the correlation of complete response to TNT with presence or absence of ctDNA
3. Describe the recurrence rate in participants with and without ctDNA after TNT
4. Characterize the correlation of ctDNA at end of TNT with recurrence free survival at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly histologically documented rectal adenocarcinoma or biopsy-proven adenoma with MRI rectum and CT chest/abdomen or PET/CT imaging consistent with stage II or III disease
* Plan is for participant to undergo standard TNT with induction chemoradiation
* Age ≥ 18 years of age

Exclusion Criteria:

* Stage I, recurrent, or metastatic rectal cancer
* Received prior therapy for this rectal cancer
* No baseline tumor biopsies with adenocarcinoma or adequate amount of tissue from biopsies available to send for SignateraTM assay development

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will consist of individuals of any gender who are 18 years of age or older. They will all have a diagnosis of stage II or III rectal adenocarcinoma or adenoma.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Detectable ctDNA at the Completion of TNT | up to 24 months after TNT
  The percentage of participants with detectable ctDNA at the completion of TNT

SECONDARY OUTCOMES:
Change in ctDNA | up to 24 months after TNT
  The change in ctDNA (continuous and categorical positive/negative) during and at the end of neoadjuvant chemoradiation and with chemotherapy will be measured. Continuous measurements will be summarized using medians and ranges. Categorical factors will be summarized using frequencies and percentages. Changes in ctDNA will be analyzed by using the Mann-Whitney U test or the Fisher's exact test for continuous or categorical variables, respectively.
Correlation of Complete Response TNT | Up to 24 months after TNT
  Correlation of complete response to TNT defined by presence or absence of ctDNA.

OTHER OUTCOMES:
The recurrence rate (local and distant) with positive ctDNA and negative ctDNA after TNT | Up to 24 months after TNT
  The recurrence rate (local and distant) is the number of participants with positive ctDNA and negative ctDNA after TNT for both participants who undergo watch and wait and those who have surgery. Non operative management (watch and wait) is offered to participants who have a complete clinical response who will comply with required surveillance. Outcomes will be recorded and described for all participants, those who underwent surgery and those who underwent non-operative management.
The correlation of ctDNA at end of TNT with relapse-free survival | After 2 years of surveillance post-TNT
  The presence or absence of ctDNA with relapse-free survival.Time to event variable will be summarized using the Kaplan-Meier method. Outcomes will be recorded and described for all patients, those who underwent surgery and those who underwent non-operative management.

CONTACTS AND LOCATIONS:
Overall Officials: Smitha Krishnamurthi, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States